CLINICAL TRIAL: NCT06251817
Title: The Wideband Acoustic Immittance Data in Thai Normal Hearing and Conductive Hearing Loss Adults
Status: Enrolling by invitation | Type: Observational
Sponsor: Khon Kaen University (Other)
Collaborators: Prince of Songkla University (Other); Chiang Mai University (Other)
Responsible Party: Principal Investigator, Nichtima Chayaopas, The collaborative Research Grants of CMU-KKU-PSU Cooperation Project, Khon Kaen University
Other Study IDs: 67/1-2-2-1-001
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Normal Hearing; Conductive Hearing Loss, Middle Ear
Keywords: wideband acoustic immittance; Normal hearing; Thai adults; Conductive hearing loss; Absorbance
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this descriptive study is to collect the wideband immittance data in Thai normal hearing and conductive hearing loss adults. The main questions it aims to answer are:

1. What is normative data of wideband acoustic immittance in Thai normal hearing adults
2. What is the wideband acoustic immittance data in Thai conductive hearing loss who have type A, AS and Ad tympanogram Participants will examine hearing tests consequently

   * pure tone audiometry
   * Tympanometry with ipsilateral acoustic reflex
   * Wideband acoustic immittance

ELIGIBILITY:
Inclusion Criteria:

Normal group

1. Thai adults (18-60 years old)
2. Pure-tone air-conduction thresholds ≤ 25 dB HL, measured at audiometric frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 and 8000 Hz and air-bone gab < 10 dBHL at frequencies 500, 1000, 2000 and 4000 Hz
3. Type A tympanogram with present ipsilateral acoustic reflex
4. No diagnosis of middle ear disease
5. No history of middle ear surgery
6. Normal finding in otoscopic examination

Conductive hearing loss group

1. Thai adults (18-60 years old)
2. Pure-tone air-conduction thresholds > 25 dB HL, measured at audiometric frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 and 8000 Hz and air-bone gab > 10 dBHL at frequencies 500, 1000, 2000 and 4000 Hz at least 2 frequencies in one ear
3. Type A, As or Ad tympanogram with absent ipsilateral acoustic reflex
4. Normal finding in otoscopic examination
5. There is an appointment for exploration middle ear within 2 months

Exclusion Criteria:

1. Have previously had middle ear surgery
2. Have an earache
3. Type B or C tympanogram
4. Volunteers who do not cooperate in audiometry test or unable to do audiometry test

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thai adults 18 to 59 years old who have normal hearing 245 participants and conductive hearing loss 45 participants
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-10-05 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Normative data of wideband acoustic immittance in Thai normal hearing adults | 3-4 months
  Normative data of wideband acoustic immittance refers to wideband absorbance at peak pressure and wideband absorbance at ambient pressure at across frequency (226 to 8000 Hz.)

SECONDARY OUTCOMES:
The wideband acoustic immittance data in Thai adults conductive hearing loss | 16-18 months
  The wideband acoustic immittance measures characteristic of conductive hearing loss with tympanogram types A, As, and Ad

CONTACTS AND LOCATIONS:
Locations (1):
- Department of otolaryngology, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided